CLINICAL TRIAL: NCT05589207
Title: Preoperative Imaging Diagnostic Evaluation Model Based on Evidence-based Pathological Diagnose Criteria for Renal Cell Carcinoma Tumor Thrombus With Inferior Vena Cava Wall Invasion
Brief Title: Predicting Model Based on Evidence-based Pathological Diagnose Criteria for RCC Tumor Thrombus With IVC Wall Invasion
Status: Recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Liu Zhuo, Attending Doctor, Peking University Third Hospital
Other Study IDs: M2022597
Record Dates: First submitted 2022-10-15; First posted 2022-10-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Carcinoma, Renal Cell; Tumor Thrombus; Neoplasm Invasiveness; Inferior Vena Cava Interruption
Keywords: Neoplasm Grading; Diagnostic Model; Preoperative Diagnosis
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasm Invasiveness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Invaded Group: Patients whose inferior vena cava vascular wall is invaded according to histopathological examination.
  Interventions: Diagnostic Test: Vascular wall invaded
- Non-invaded group: Patients whose inferior vena cava vascular wall is not invaded according to histopathological examination.

INTERVENTIONS:
Diagnostic Test: Vascular wall invaded — Inferior vena cava vascular wall is invaded according to pathologic examination on the postoperative tumor thrombus/ vascular wall specimen.
  Groups: Invaded Group

SUMMARY:
The goal of this observational study is to establish a preoperative imaging diagnostic model which highly consistent with the histopathological examinations, as well as a accurate and systematic pathological grading standard of inferior vena cava (IVC) vascular wall invasion in renal cell carcinoma (RCC) with tumor thrombus invading vascular wall.The main questions it aims to answer are:

* To establish a preoperative imaging diagnostic model which highly consistent with the histopathological examinations.
* To determine what impact does different vascular wall layer invasion make on the long-term prognosis in RCC with IVC tumor thrombus;
* To determine which layer invasion according to pathological examination make sense to clinical treatment (can significantly affect prognosis); Participants with IVC vascular wall invasion/ non-invasion are divided into experimental group (invaded group) or control group (non-invaded group) respectively according to pathological examinations, in order to establish a prospective cohort with three-year follow-up. The pathological characteristics of local recurrence and poor prognosis are summarized, and postoperative pathological diagnostic criteria of IVC vascular wall invasion and established. The local recurrence and distant recurrence outcomes are compared between experiment group and control group, in order to analyze the long-term influence of vascular wall invasion. Then the preoperative imaging diagnostic evaluation model will be established.

DETAILED DESCRIPTION:
Radical nephrectomy and thrombectomy are essential surgical treatments for renal cell carcinoma (RCC) with inferior vena cava (IVC) tumor thrombus. IVC vascular wall invasion leads to higher recurrence risk and worse long-term prognosis. The diagnosis and treatment of RCC tumor thrombus with IVC vascular wall invaded are affected by prominent difficulties: First, there is a lack of the preoperative diagnostic evaluation system consisting to the postoperative histopathological examinations, which is regarded as the gold standard of vascular wall invasion, therefore hinders the development of the neoadjuvant therapy strategy and surgery plan; Besides, the pathological diagnostic criteria of IVC vascular wall adhesion or invasion is inconsistent among different centers, an accurate and systematic criteria is needed.

This study consecutively includes patients admitted in Peking University Third Hospital between January 2023 to January 2026, who were diagnosed with primary renal cell carcinoma with IVC tumor thrombus with/without vascular wall invasion, and accepted radical nephrectomy and at least one IVC thrombectomy (including IVC incision only, IVC partial resection, IVC diagonal resection, and IVC segmental resection). The patients with IVC vascular wall invasion/ non-invasion are divided into experimental group (invaded group) or control group (non-invaded group) respectively according to pathological examinations, in order to establish a prospective cohort with three-year follow-up. For the invaded group, micro invasion subgroup and tumor thrombus capsule subgroup analysis are conducted. The pathological characteristics of local recurrence and poor prognosis are summarized, and postoperative pathological diagnostic criteria of IVC vascular wall invasion and established. The local recurrence and distant recurrences outcomes are compared between experiment group and control group, in order to analyze the long-term influence of vascular wall invasion. Then the preoperative imaging diagnostic evaluation model were established: re-diagnose patients in two groups according to the established pathological diagnostic criteria, and divide them into truly-invaded group and truly-non-invaded group. Analyzing the preoperative abdominal ultrasound scan, contrast-enhanced ultrasonography, computed tomography (CT) and magnetic resonance imaging (MRI), thus explore the imaging characteristics of vascular wall invasion and establish the preoperative diagnostic model. This study aims at establish a preoperative imaging diagnostic model which highly consistent with the histopathological examinations, as well as a accurate and systematic pathological grading standard of IVC vascular wall invasion, therefore contribute to the development of a more accurate and effective preoperative treatment strategy and surgery plan.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years of age;
* Accepted abdominal ultrasonography, contrast-induced ultrasonography, enhanced CT and MRI before the surgery;
* Diagnosis of primary renal cell carcinoma with tumor thrombus before and during the surgery;
* Received radical nephrectomy and at least one kind of thrombectomy (including IVC incision only, IVC partial resection, IVC diagonal resection, and IVC segmental resection)
* Can tolerate the surgery;
* Eastern Cooperative Oncology Group Performance Status Scale (ECOG-PS) 0~2;
* No previous history of malignant tumor;
* Willing to return for required follow-up visits

Exclusion Criteria:

* Failed to receive standard nephrectomy for any reason;
* Attached other addition operations in the surgery;
* Received neoadjuvant treatment before the surgery;
* Experience any other conditions that may affect the curative effect (e.g. active tuberculosis, autoimmune disease, or oral glucocorticoids treatment);
* Experience serious consequences or death due to anesthesia accident during operation;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The groups of cohort will be selected from inhospital patients in Peking University Third Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 232 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | From date of randomization until the date of lost follow-up or date of death from any cause, whichever came first, assessed up to 120 months
  The duration from the date of diagnosis to death or last follow-up, with no restriction on the cause of death.

SECONDARY OUTCOMES:
Clinical manifestation | From the clinical diagnosis until the surgery, an average of 3 weeks
  Clinical manifestation related to the renal carcinoma
Mayo classification | The time once the preoperative imaging is assessed, up to 1 weeks.
  A universal grading system for renal tumor thrombus.
Primary tumor diameter | The time once the preoperative imaging is assessed, up to 1 weeks.
  Diameter of the primary tumor.
Preoperative tumor node metastasis (TNM) stage | The time once the preoperative imaging is assessed, up to 1 weeks.
  TNM stage according to the preoperative imaging.
IVC residual blood flow | The time once the preoperative imaging is assessed, up to 1 weeks.
  Inferior vena cava residual blood flow according to ultrasonography.
IVC vascular wall continuity | The time once the preoperative imaging is assessed, up to 1 weeks.
  Inferior vena cava vascular wall continuity according to ultrasonography.
IVC complete occlusion | The time once the preoperative imaging is assessed, up to 1 weeks.
  Whether the inferior vena cava is completely occluded according to ultrasonography.
IVC enhanced synchronization with tumor thrombus | The time once the preoperative imaging is assessed, up to 1 weeks.
  Whether the inferior vena cava enhanced synchronization with tumor thrombus according to ultrasonography.
Tumor thrombus move when breathe | The time once the preoperative imaging is assessed, up to 1 weeks.
  Whether the tumor thrombus move when breathe according to ultrasonography.
Maximum IVC anterior-posterior (AP) diameter | The time once the preoperative imaging was assessed, up to 1 weeks.
  Maximum inferior vena cava anterior-posterior diameter according to CT/ MRI.
Maximum coronal IVC diameter | The time once the preoperative imaging is assessed, up to 1 weeks.
  Maximun coronal inferior vena cava diameter according to CT/ MRI.
Maximum IVC AP diameter at the Rvo | The time once the preoperative imaging is assessed, up to 1 weeks.
  Maximum inferior vena cava anterior-posterior diameter at the renal vein ostium according to CT/ MRI.
Maximum coronal IVC diameter at the Rvo | The time once the preoperative imaging is assessed, up to 1 weeks.
  Maximun coronal inferior vena cava diameter at the renal vein ostium according to CT/ MRI.
Bland thrombus | The time once the preoperative imaging is assessed, up to 1 weeks.
  The presence of bland thrombus in inferior vena cava according to CT/ MRI.
growing against the direction of venous return (GADVR) | The time once the preoperative imaging is assessed, up to 1 weeks.
  The presence of tumor thrombus growing against the direction of venous return according to CT/ MRI.
Surgery approach | The time once the surgery finished, an average of 10 days.
  Radical nephrectomy and at least one kind of IVC thrombectomy (including IVC incision only, IVC partial resection, IVC diagonal resection, and IVC segmental resection)
Surgery time | The time once the surgery finished, an average of 10 days.
  Surgery time
Blood loss | The time once the surgery finished, an average of 10 days.
  Blood loss during surgery
Histological type | The time once the pathological specimen is assessed, up to 1 weeks.
  Histological type of the tumor according to pathological examination.
Postoperative TNM stage | The time once the pathological specimen is assessed, up to 1 weeks.
  TNM stage according to pathological examination.
Invaded vascular wall layer | The time once the pathological specimen is assessed, up to 1 weeks.
  The deepest Inferior vane cava vascular wall layer the tumor thrombus invaded.
Comorbidity occurence | From the end of surgery until discharge, up to 3 weeks.
  The comorbidity occurence after surgery.
Recurrence free survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 120 months
  The duration from the date of diagnosis to death, last follow-up, or cancer recurrence.
Tumor metastasis | Through study completion, an average of 3 year.
  Location and time that the metastasis occurs.

CONTACTS AND LOCATIONS:
Overall Officials: Zhuo Liu, MD, Study Director — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Adams LC, Ralla B, Bender YY, Bressem K, Hamm B, Busch J, Fuller F, Makowski MR. Renal cell carcinoma with venous extension: prediction of inferior vena cava wall invasion by MRI. Cancer Imaging. 2018 May 3;18(1):17. doi: 10.1186/s40644-018-0150-z. PMID 29724245
- [Background] Ingels A, Campi R, Capitanio U, Amparore D, Bertolo R, Carbonara U, Erdem S, Kara O, Klatte T, Kriegmair MC, Marchioni M, Mir MC, Ouzaid I, Pavan N, Pecoraro A, Roussel E, de la Taille A. Complementary roles of surgery and systemic treatment in clear cell renal cell carcinoma. Nat Rev Urol. 2022 Jul;19(7):391-418. doi: 10.1038/s41585-022-00592-3. Epub 2022 May 11. PMID 35546184
- [Background] Labbate C, Hatogai K, Werntz R, Stadler WM, Steinberg GD, Eggener S, Sweis RF. Complete response of renal cell carcinoma vena cava tumor thrombus to neoadjuvant immunotherapy. J Immunother Cancer. 2019 Mar 11;7(1):66. doi: 10.1186/s40425-019-0546-8. PMID 30857555
- [Background] Shi T, Huang Q, Liu K, Du S, Fan Y, Yang L, Peng C, Shen D, Wang Z, Gao Y, Gu L, Niu S, Ai Q, Li H, Liu F, Li Q, Wang H, Guo A, Fu B, Yang X, Zhang X, Wang D, Wang D, Guo H, Li H, Olivero A, Fam XI, Ma X, Wang B, Zhang X. Robot-assisted Cavectomy Versus Thrombectomy for Level II Inferior Vena Cava Thrombus: Decision-making Scheme and Multi-institutional Analysis. Eur Urol. 2020 Oct;78(4):592-602. doi: 10.1016/j.eururo.2020.03.020. Epub 2020 Apr 15. PMID 32305170
- [Background] Liu Z, Zhao X, Zhang HX, Li LW, Tang SY, Wang GL, Zhang SD, Wang SM, Ma LL, Tian XJ. Surgical complexity and prognostic outcome of small volume renal cell carcinoma with high-level venous tumor thrombus and large volume renal cell carcinoma with low-level thrombus. Chin Med J (Engl). 2019 Aug 5;132(15):1780-1787. doi: 10.1097/CM9.0000000000000352. PMID 31306232
- [Background] Rodriguez Faba O, Linares E, Tilki D, Capitanio U, Evans CP, Montorsi F, Martinez-Salamanca JI, Libertino J, Gontero P, Palou J. Impact of Microscopic Wall Invasion of the Renal Vein or Inferior Vena Cava on Cancer-specific Survival in Patients with Renal Cell Carcinoma and Tumor Thrombus: A Multi-institutional Analysis from the International Renal Cell Carcinoma-Venous Thrombus Consortium. Eur Urol Focus. 2018 Apr;4(3):435-441. doi: 10.1016/j.euf.2017.01.009. Epub 2017 Feb 9. PMID 28753848
- [Background] Lardas M, Stewart F, Scrimgeour D, Hofmann F, Marconi L, Dabestani S, Bex A, Volpe A, Canfield SE, Staehler M, Hora M, Powles T, Merseburger AS, Kuczyk MA, Bensalah K, Mulders PF, Ljungberg B, Lam TB. Systematic Review of Surgical Management of Nonmetastatic Renal Cell Carcinoma with Vena Caval Thrombus. Eur Urol. 2016 Aug;70(2):265-80. doi: 10.1016/j.eururo.2015.11.034. Epub 2015 Dec 23. PMID 26707869
- [Background] Wagner B, Patard JJ, Mejean A, Bensalah K, Verhoest G, Zigeuner R, Ficarra V, Tostain J, Mulders P, Chautard D, Descotes JL, de la Taille A, Salomon L, Prayer-Galetti T, Cindolo L, Valeri A, Meyer N, Jacqmin D, Lang H. Prognostic value of renal vein and inferior vena cava involvement in renal cell carcinoma. Eur Urol. 2009 Feb;55(2):452-9. doi: 10.1016/j.eururo.2008.07.053. Epub 2008 Aug 5. PMID 18692951
- [Background] Liu Z, Li L, Hong P, Zhu G, Tang S, Zhao X, Zhang Q, Wang G, He W, Zhang H, Xue H, Cui L, Ge H, Jiang J, Zhang S, Cao F, Yan J, Ma F, Liu C, Ma L, Wang S. A Predictive Model for Tumor Invasion of the Inferior Vena Cava Wall Using Multimodal Imaging in Patients with Renal Cell Carcinoma and Inferior Vena Cava Tumor Thrombus. Biomed Res Int. 2020 Oct 6;2020:9530618. doi: 10.1155/2020/9530618. eCollection 2020. PMID 33083491
- [Background] Wang BS, Li YZ, Fang YY, Zhang SD, Ma LL. Imaging predictors for assessment of inferior vena cava wall invasion in patients with renal cell carcinoma and inferior vena cava tumor thrombus: a retrospective study. Chin Med J (Engl). 2020 Sep 5;133(17):2078-2083. doi: 10.1097/CM9.0000000000000828. PMID 32898352
- [Background] Li QY, Li N, Huang QB, Luo YK, Wang BJ, Guo AT, Ma X, Zhang X, Tang J. Contrast-enhanced ultrasound in detecting wall invasion and differentiating bland from tumor thrombus during robot-assisted inferior vena cava thrombectomy for renal cell carcinoma. Cancer Imaging. 2019 Dec 2;19(1):79. doi: 10.1186/s40644-019-0265-x. PMID 31791422
- [Background] Sun Z, Cui Y, Xu C, Yu Y, Han C, Liu X, Lin Z, Wang X, Li C, Zhang X, Wang X. Preoperative Prediction of Inferior Vena Cava Wall Invasion of Tumor Thrombus in Renal Cell Carcinoma: Radiomics Models Based on Magnetic Resonance Imaging. Front Oncol. 2022 Jun 6;12:863534. doi: 10.3389/fonc.2022.863534. eCollection 2022. PMID 35734586
- [Background] Ueki H, Terakawa T, Ueno Y, Sofue K, Horii S, Okamura Y, Bando Y, Hara T, Furukawa J, Harada K, Hinata N, Nakano Y, Murakami T, Fujisawa M. Efficacy of preoperative cine magnetic resonance imaging in evaluation of adhesion of renal cancer thrombus to inferior vena cava wall. J Vasc Surg Venous Lymphat Disord. 2022 Jul;10(4):908-915. doi: 10.1016/j.jvsv.2022.02.016. Epub 2022 Mar 18. PMID 35314389
- [Background] Hirono M, Kobayashi M, Tsushima T, Obara W, Shinohara N, Ito K, Eto M, Takayama T, Fujii Y, Nishikido M, Kimura G, Kishida T, Takahashi M, Miyao N, Naya Y, Abe T, Fujioka T, Ito K, Naito S; Members of the Japanese Society of Renal Cancer. Impacts of clinicopathologic and operative factors on short-term and long-term survival in renal cell carcinoma with venous tumor thrombus extension: a multi-institutional retrospective study in Japan. BMC Cancer. 2013 Oct 2;13:447. doi: 10.1186/1471-2407-13-447. PMID 24083566
- [Background] Liu Z, Zhang Q, Zhao X, Zhu G, Tang S, Hong P, Ge L, Zhang S, Wang G, Tian X, Zhang H, Liu C, Ma L. Inferior vena cava interruption in renal cell carcinoma with tumor thrombus: surgical strategy and perioperative results. BMC Surg. 2021 Nov 21;21(1):402. doi: 10.1186/s12893-021-01400-2. PMID 34802447
- [Background] Abaza R. Initial series of robotic radical nephrectomy with vena caval tumor thrombectomy. Eur Urol. 2011 Apr;59(4):652-6. doi: 10.1016/j.eururo.2010.08.038. Epub 2010 Sep 16. PMID 20846783
- [Background] Wang B, Huang Q, Liu K, Fan Y, Peng C, Gu L, Shi T, Zhang P, Chen W, Du S, Niu S, Liu R, Zhao G, Li Q, Xiao C, Wang R, Li S, Wang M, Liu F, Wang H, Li H, Ma X, Zhang X. Robot-assisted Level III-IV Inferior Vena Cava Thrombectomy: Initial Series with Step-by-step Procedures and 1-yr Outcomes. Eur Urol. 2020 Jul;78(1):77-86. doi: 10.1016/j.eururo.2019.04.019. Epub 2019 May 16. PMID 31103390
- [Background] Liu Z, Li Y, Zhao X, Ge L, Zhu G, Hong P, Tang S, Zhang S, Tian X, Wang S, Liu C, Zhang H, Ma L. Renal cell carcinoma with tumor thrombus growing against the direction of venous return: an indicator of complicated surgery and poor prognosis. BMC Surg. 2021 Dec 28;21(1):443. doi: 10.1186/s12893-021-01448-0. PMID 34963464
- [Background] Bocardo Fajardo G, Arellano Ganan R, Gonzalez Lopez L, Fernandez Gonzalez I, Blanco Gonzalez J, Garrido Abad P, Coloma del Peso A, Pereira Sanz I. [Prognostic significance of the microscopic invasion of the renal vein wall in renal cell cancer]. Arch Esp Urol. 2009 Oct;62(8):630-8. doi: 10.4321/s0004-06142009000800004. Spanish. PMID 19893136
- [Background] Lang H, Lindner V, Saussine C, Havel D, Faure F, Jacqmin D. Microscopic venous invasion: a prognostic factor in renal cell carcinoma. Eur Urol. 2000 Nov;38(5):600-5. doi: 10.1159/000020338. PMID 11096243
- [Background] Lakatos E. Sample sizes based on the log-rank statistic in complex clinical trials. Biometrics. 1988 Mar;44(1):229-41. PMID 3358991
- [Background] Lakatos E. Designing complex group sequential survival trials. Stat Med. 2002 Jul 30;21(14):1969-89. doi: 10.1002/sim.1193. PMID 12111882